CLINICAL TRIAL: NCT00000737
Title: A Phase I/II Study to Evaluate Single Agent and Combination Therapy With Megestrol Acetate and Dronabinol for the Treatment of HIV-Wasting Syndrome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Roxane Laboratories (Industry); Bristol-Myers Squibb (Industry)
Masking: None | Purpose: Treatment
Other Study IDs: DATRI 004
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2008-08-25 (Estimated); Status verified 1994-01

CONDITIONS: Cachexia; HIV Infections; HIV Wasting Syndrome
Keywords: Weight Loss; Megestrol; Cachexia; Eating Disorders; Tetrahydrocannabinol; Appetite
MeSH Terms: conditions — Cachexia; HIV Infections; HIV Wasting Syndrome; Weight Loss; Feeding and Eating Disorders | interventions — Dronabinol; Megestrol Acetate

INTERVENTIONS:
Drug: Dronabinol
Drug: Megestrol acetate

SUMMARY:
To obtain data on the safety of administering megestrol acetate and dronabinol as single agents or in combination to patients with human immunodeficiency virus (HIV)-wasting syndrome. To obtain preliminary data on the efficacy of single agent and combination therapy with megestrol acetate and dronabinol with regard to weight gain, appetite increase and quality of life in this patient population. To obtain steady-state pharmacokinetics data when megestrol acetate and dronabinol are administered as single agents and in combination.

HIV-wasting syndrome, which is characterized by severely debilitating anorexia and weight loss, is of particular concern because it can exacerbate the primary illness and is associated with a poor prognosis. Attempts at maintaining body mass through the use of megestrol acetate and dronabinol, two anti-cachectic drugs, may prolong survival.

DETAILED DESCRIPTION:
HIV-wasting syndrome, which is characterized by severely debilitating anorexia and weight loss, is of particular concern because it can exacerbate the primary illness and is associated with a poor prognosis. Attempts at maintaining body mass through the use of megestrol acetate and dronabinol, two anti-cachectic drugs, may prolong survival.

Fifty-six patients are randomized to one of four treatment arms, as follows: high-dose megestrol acetate alone; dronabinol alone; high-dose megestrol acetate combined with dronabinol; or low-dose megestrol acetate combined with dronabinol. Treatment continues for 12 weeks. Patients are evaluated for toxicity, preliminary evidence of response (e.g., weight gain), and steady-state pharmacokinetics of drug therapies.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Zidovudine (AZT), didanosine (ddI), and dideoxycytidine (ddC). If initiating new antiretroviral therapy, patient must have been on a stable dose for at least 4 weeks prior to study entry.
* Maintenance or suppressive therapy with any of the following, provided patient has been on a stable dose for at least 1 week prior to study entry:
* Ganciclovir or foscarnet for CMV retinitis.
* Fluconazole, amphotericin B, or flucytosine for cryptococcosis.
* Amphotericin B for disseminated histoplasmosis.
* Pyrimethamine, sulfadiazine, dapsone, or clindamycin for toxoplasmosis.
* Amikacin, clarithromycin, clofazimine, ethambutol, ciprofloxacin, or rifampin for disseminated Mycobacterium avium complex.
* Isoniazid, rifampin, ethambutol, or pyrazinamide for M. tuberculosis.
* Any of the following provided patient is on a stable dose for at least 1 week prior to study entry:
* Trimethoprim-sulfamethoxazole, aerosolized pentamidine, or dapsone for Pneumocystis carinii prophylaxis.
* Clotrimazole troches, nystatin suspension, ketoconazole, or fluconazole for oral candidiasis.
* Oral acyclovir for mucocutaneous herpes simplex.
* Narcotic analgesics, tranquilizers, sedative-hypnotics, or anticholinergic agents provided patient is on a stable dose for at least 1 week prior to study entry.

Patients must have:

* HIV infection.
* HIV-wasting syndrome and anorexia.
* Life expectancy of at least 4 months.
* Ability to tolerate oral therapy, feed themselves, and have access to as much food as they desire with no dietary restrictions.

Prior Medication:

Allowed:

* Prior zidovudine (AZT), didanosine (ddI), and dideoxycytidine (ddC).
* Prior maintenance or suppressive therapy for certain opportunistic infections, as follows:
* Ganciclovir or foscarnet for CMV retinitis.
* Fluconazole, amphotericin B, or flucytosine for cryptococcosis.
* Amphotericin B for disseminated histoplasmosis.
* Pyrimethamine, sulfadiazine, dapsone, or clindamycin for toxoplasmosis.
* Amikacin, clarithromycin, clofazimine, ethambutol, ciprofloxacin, or rifampin for disseminated Mycobacterium avium complex.
* Isoniazid, rifampin, ethambutol, or pyrazinamide for M. tuberculosis.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Major, acute opportunistic infections.
* Active neoplasms other than Kaposi's sarcoma or localized skin carcinoma.
* Diabetes, congestive heart failure, clinical ascites, or uncontrolled hypertension.
* Persistent grade 3/4 diarrhea.
* Impaired oral intake, such as occurs with Candida esophagitis or severe mouth ulcers.
* Clinically significant cardiac arrhythmias.
* Requirement for anticonvulsants for seizure disorder.

Concurrent Medication:

Excluded:

* Marijuana use.
* Anabolic steroids.
* Anticonvulsants for seizure disorders.
* Alcohol or barbiturates.

Patients with the following prior conditions are excluded:

* Diagnosis of a major, acute opportunistic infection within 2 months prior to study entry.
* Hospitalization within 2 weeks prior to study entry.
* History of hypersensitivity reactions to megestrol acetate, dronabinol, or sesame oil (a component of the dronabinol capsules).
* History of thromboembolic events.
* History of psychiatric disorder other than depression.

Prior Medication:

Excluded:

* Prior dronabinol.
* Megestrol acetate within 2 months prior to study entry.
* Marijuana within 1 month prior to study entry.
* Anabolic steroids within 3 months prior to study entry.

Current drug or alcohol abuse (patients with a history of occasional marijuana use are eligible provided they have abstained from its use for 1 month prior to study entry and agree to refrain from marijuana use for the study period).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56

CONTACTS AND LOCATIONS:
Overall Officials: Galetto G, Study Chair; Egorin M, Study Chair
Locations (9):
- United States (9):
  - Denver Public Health Dept, Denver, Colorado
  - Univ of Illinois, Chicago, Illinois
  - Univ of Kansas School of Medicine, Wichita, Kansas
  - Tulane Univ Med School, New Orleans, Louisiana
  - Univ of Maryland at Baltimore / Veterans Adm, Baltimore, Maryland
  - Washington Univ, St Louis, Missouri
  - SUNY / Health Sciences Ctr at Brooklyn, Brooklyn, New York
  - Portland Veterans Adm Med Ctr / Rsch & Education Grp, Portland, Oregon
  - Univ of Rhode Island / College of Pharmacy, Providence, Rhode Island

REFERENCES:
- [Background] Timpone JG, Wright DJ, Li N, Egorin MJ, Enama ME, Mayers J, Galetto G. The safety and pharmacokinetics of single-agent and combination therapy with megestrol acetate and dronabinol for the treatment of HIV wasting syndrome. The DATRI 004 Study Group. Division of AIDS Treatment Research Initiative. AIDS Res Hum Retroviruses. 1997 Mar 1;13(4):305-15. doi: 10.1089/aid.1997.13.305. PMID 9071430